CLINICAL TRIAL: NCT05410756
Title: Relationship Between Dysphonia And Anxiety In Fibromyalgia Syndrome
Brief Title: Relationship Between Dysphonia And Anxiety In Fibromyalgia
Status: Completed | Type: Observational
Sponsor: Umraniye Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Özlem Kaleoğlu Aslan, Director, Umraniye Education and Research Hospital
Other Study IDs: B.10.1.THK.4.34.H.GP.0.01
Record Dates: First submitted 2022-06-04; First posted 2022-06-08 (Actual); Last update posted 2022-06-15 (Actual); Status verified 2022-06

CONDITIONS: Dysphonia; Fibromyalgia; Anxiety Disorders
Keywords: anxiety; fibromyalgia; dysphonia
MeSH Terms: conditions — Dysphonia; Fibromyalgia; Anxiety Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- FIBROMYALGIA GROUP: Patients diagnosed with Fibromyalgia Syndrome (n=25) who volunteered to be undergone voice analysis.
  Interventions: Diagnostic Test: Assessment of Voice Quality and Function
- HEALTHY CONTROL GROUP: Healthy volunteers (n=25) without any chronic disease not under any medication volunteered to be undergone voice analysis.
  Interventions: Diagnostic Test: Assessment of Voice Quality and Function

INTERVENTIONS:
Diagnostic Test: Assessment of Voice Quality and Function — An acoustic voice analysis (fundamental frequency (F0), jitter, shimmer, noise to harmonic ratio (NHR), harmonic to noise ratio (HNR)) and an aerodynamic analysis (maximal phonation time (MPT)) were performed by an experienced otolaryngologist specialized in voice disorders for evaluation of objective voice quality and function. These analyses were performed on all the volunteers from both groups, and the results obtained were compared between the groups.

SUMMARY:
Our aim in conducting this study is to determine the relationship between voice disorders and anxiety in patients with fibromyalgia syndrome (FS).

DETAILED DESCRIPTION:
This case controlled study was performed at the Physical Medicine and Rehabilitation outpatient clinic between April 2022 and June 2022. 25 patients who were diagnosed with FS according to the 2010 American College of Rheumatology (ACR) criteria were included in the study. For the control group 25 healthy volunteers with no previous chronic disease history were included . The investigators planed to investigate the relationship between the anxiety level of the FS patients and dysphonia. Thus an acoustic voice analysis (fundamental frequency (F0), jitter, shimmer, noise to harmonic ratio (NHR), harmonic to noise ratio (HNR)) and an aerodynamic analysis (maximal phonation time (MPT)) were performed by an experienced otolaryngologist specialized in voice disorders for evaluation of objective voice quality and function. These analyses were performed on all the volunteers from both groups, and the results obtained were compared between the groups.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Fibromyalgia syndrome for at least 1 year
* Minimum VAS score of 3

Exclusion Criteria:

* Patients with diabetes mellitus,
* other rheumatological diseases,
* malignancies,
* connective tissue disorders
* neuromuscular diseases and
* hereditary diseases.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 25 patients diagnosed with fibromyalgia syndrome
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
Beck Anxiety Questionary Score | at the start of the study
  Measuring The Anxiety level, It is scored between 0-63. The greater the score the greater the anxiety level of the subject.
Visual Analogue Scale (VAS) Score | at the start of the study
  Visual Analogue Scale is used to measure the pain level of the subjects. It is scored between 0 to 10. Greater score corresponds to greater pain sensation.

CONTACTS AND LOCATIONS:
Overall Officials: Özlem Aslan, Principal Investigator — Umraniye Education and Research Hospital
Locations (1):
- Umraniye Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No